CLINICAL TRIAL: NCT01947985
Title: A Pharmacoepidemiological Study of Rivaroxaban Use and Potential Adverse Outcomes in Routine Clinical Pratice in the Netherlands.
Brief Title: Study of Rivaroxaban Use and Potential Adverse Outcomes in Routine Clinical Pratice (Netherlands)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16646; EUPAS11141 (Registry Identifier: ENCEPP)
Record Dates: First submitted 2013-09-11; First posted 2013-09-23 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation; Acute Coronary Syndrome
Keywords: Rivaroxaban; Stroke Prevention in Atrial Fibrillation; Anticoagulants; Hematologic Agents; Therapeutic Uses; Observational; Venous Thromboembolism; Secondary Prevention of Acute Coronary Syndrome; Intracranial Hemorrhages; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation; Acute Coronary Syndrome; Venous Thromboembolism; Intracranial Hemorrhages; Gastrointestinal Hemorrhage | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rivaroxoban: Patients who have been prescribed Rivaroxaban for the first time
  Interventions: Drug: Rivaroxoban (Xarelto, Bay59-7939)
- Standard of care: Patients who have been prescribed standard of care for the first time
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Rivaroxoban (Xarelto, Bay59-7939) — The treatment of deep vein thrombosis (DVT) or pulmonary embolism (PE), and prevention of recurrent DVT and PE in adult patients (15 mg rivaroxaban twice daily [bid] for 3 weeks, then 15 mg or 20 mg once daily [od], tablets).
  The prevention of stroke and systemic embolism in adult patients with non-valvular atrial fibrillation (stroke prevention in atrial fibrillation [SPAF]) with one or more risk factors (20 mg rivaroxaban [od], tablets).
  The prevention of venous thromboembolism (VTE) in adult patients undergoing elective hip or knee replacement surgery (recommended dose: 10 mg rivaroxaban [od] tablets for 35 days following hip replacement surgery and 14 days following knee replacement surgery).
  Co-administered with acetylsalicylic acid (ASA) alone or with ASA plus clopidogrel or ticlopidine, for the prevention of atherothrombotic events in adult patients after an acute coronary syndrome (ACS) with elevated cardiac biomarkers (recommended dose 2.5 mg rivaroxaban tablets [bid]).
  Groups: Rivaroxoban
Drug: Standard of care — For DVT/PE treatment and SPAF, standard of care is treatment with the most widely used vitamin K antagonist, phenprocoumon, and for the secondary prevention of ACS, standard of care is antiplatelet drug(s) such as low-dose acetylsalicylic acid, clopidogrel, dipyridamole, prasugrel, ticlopidine and ticagrelor.
  Groups: Standard of care

SUMMARY:
This prospective cohort study will provide information about: characteristics of Rivaroxaban use in patients who are prescribed Rivaroxaban for the first time compared to patients who are prescribed Acenocoumarol for the first time, the occurrence of intracranial haemorrhage, gastrointestinal and urogenital bleeding, and the occurrence of non-infective liver disease.

ELIGIBILITY:
Inclusion Criteria:

* All male and female patients who have been prescribed for the first time either Rivaroxaban or standard of care from the date of market authorization of rivaroxaban to Dec 31, 2017

Exclusion Criteria:

* Patients who have any record of being dispensed their index drug in the year before index date (i.e. cohort entry), or who qualify for both cohorts on the same day will be excluded

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 2 years and above who have been registered in the PHARMO database for at least 1 year before the index date.
Sampling Method: Non-Probability Sample
Enrollment: 208958 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of demographic and clinical characteristics of patients who are prescribed oral rivaroxaban for the first time in comparison with those who are prescribed standard of care for the first time | up to 8 years
  Age and sex distribution at index date Proportion of patients defined as naïve, non-naïve, recent switchers and distant switchers Type and estimated duration of other anticoagulant use among the non-naïve group and for all patients Number of pregnancies and pregnancy outcomes' Use of specific prescribed medications confirming ACS indication Use of other prescribed medications Renal disease based on in- and outpatient diagnoses Hospital admissions for bleeding Healthcare utilization (e.g. number of hospital admissions). Smoking status Body mass index (BMI)
Characteristics of rivaroxaban use in comparison with standard of care | up to 8 years
  Estimated dose of index drug at index date and estimated duration of treatment Where available, the diagnosis associated with the prescribing of the index drug (where not available, estimated dose and duration of index drug will be used as a proxy for the associated diagnosis among rivaroxaban users) Dispensed amount (can be used to estimate duration of treatment)
Safety: occurrence of intracranial haemorrhage leading to hospitalization among users of rivaroxaban in comparison with individuals receiving current standard of care | up to 8 years
  Cases of intracranial haemorrhage will be identified in patients admitted to the hospital that meet the criteria for one of the three following categories:
  Incident cases of intracerebral haemorrhage Incident cases of subarachnoid haemorrhage incident cases of epidural, dural, subdural and arachnoid haemorrhage Potential cases will be identified by hospital discharge diagnoses
Safety: occurrence of gastrointestinal bleeding leading to hospitalization among users of rivaroxaban in comparison with individuals receiving current standard of care | up to 8 years
  A patient will have to meet the following criteria to be considered a case of gastrointestinal bleeding:
  The specific site of bleeding originating in the upper or lower gastrointestinal tract or, more specifically, in the oesophagus, stomach, duodenum, jejunum, ileum, colon or rectum.
  For upper gastrointestinal bleeding, the lesion type being erosion, gastritis, duodenitis or peptic (gastric or duodenal) ulcer.
  The lesion type being NOT related to cancer. Cases will be identified by hospital discharge diagnoses (ICD-9-CM).
Safety: occurrence urogenital bleeding leading to hospitalization among users of rivaroxaban in comparison with individuals receiving current standard of care | up to 8 years
  A patient will have to be admitted to the hospital for urogenital bleeding, i.e. the specific site of bleeding originating in the urogenital tract.
  Cases will be identified by hospital discharge diagnoses (ICD-9-CM).

SECONDARY OUTCOMES:
Safety: occurrence of bleeding events leading to hospitalization not specified as primary safety outcomes ("other bleeding") in individuals receiving rivaroxaban, in comparison with those receiving current standard of care | up to 8 years
  A patient will have to meet the following criteria to be considered a case of "other bleeding":
  Admitted to hospital with a bleeding event occurring before hospitalization (i.e. excluding inhospital bleeding events).
  Cases will be identified by hospital discharge diagnoses (ICD-9-CM).
Safety: occurrence of non-infective liver disease leading to hospitalization in individuals receiving rivaroxaban in comparison with those receiving current standard of care | up to 8 years
  A patient will have to meet both of the following criteria to be considered a case of non-infective liver disease:
  The patient having been admitted to hospital with acute liver injury. Free of cancer, other liver disease (including infectious hepatitis, chronic liver disease etc.), gallbladder or pancreatic disease and alcoholism.
Effectiveness: occurrence of deep vein thrombosis (DVT) or pulmonary embolism (PE) in individuals receiving rivaroxaban in comparison with those receiving current standard of care | up to 8 years
  A patient will have to meet the following criteria to be considered a case of DVT or PE:
  The patient having been admitted to hospital with a diagnosis of DVT or PE or having a DVT or PE diagnosis documented in the general practitioner database.
Effectiveness: occurrence of Ischaemic stroke in individuals receiving rivaroxaban in comparison with those receiving current standard of care | up to 8 years
  A patient will have to meet the following criteria to be considered a case of ischaemic stroke: the patient having been admitted to hospital with a diagnosis of ischaemic stroke.
Effectiveness: occurrence acute myocardial infarction (MI) in individuals receiving rivaroxaban in comparison with those receiving current standard of care | up to 8 years
  A patient will have to meet the following criteria to be considered a case of MI: the patient having been admitted to hospital with a diagnosis of MI.
All-cause mortality as well as cause-specific mortality | up to 8 years
  Date of death as registered in the different databases (GP, pharmacy, hospital deaths) and confirmed through linkage with the Dutch central bureau of genealogy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Netherlands

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/